CLINICAL TRIAL: NCT04951037
Title: Producing a Fully Asynchronous Online Savvy Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Fayron Epps, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000749; 3P30AG064200-02S1 (NIH)
Record Dates: First submitted 2021-06-28; First posted 2021-07-06 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Dementia
Keywords: Dementia caregiver
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fully Asynchronous Online Savvy Program (Experimental): Family caregivers of PLWD taking part in a fully asynchronous online caregiver education program.
  Interventions: Behavioral: Fully Asynchronous Online Savvy Program

INTERVENTIONS:
Behavioral: Fully Asynchronous Online Savvy Program — The intervention is a fully online, self-administered psychoeducational program designed to enhance caregiver mastery for family and friends providing unpaid care for living with Alzheimer's and similar dementia disorders. Participants will be asked to engage with a fully online version of Tele-Savvy for 42 days.
  Participants will receive a series of daily video lessons related to caregiving. These lessons are generally 8-15 minutes in length and are emailed to participants. Participants can watch the lessons whenever and as often as they wish over the course of the study. There will also be self-guided learning strategies and exercises to accomplish skill and mastery related to the caregiving role. The lessons cover a variety of topics including:
  * Facts about dementing Illnesses
  * Caregiving Strategies - guiding the person through days that are as safe, calm, and pleasant as possible
  * Self-Care for the Caregiver
  Other Names: Tele-Savvy

SUMMARY:
This is a pilot/feasibility study to develop and test a fully online, self-administered psychoeducation program to enhance the caregiving mastery of family and friends who provide unpaid care for persons living with Alzheimer's and similar dementia disorders (PLWD).

DETAILED DESCRIPTION:
This study seeks to develop and test a fully online, self-administered psychoeducation program to enhance the caregiving mastery of family and friends who provide unpaid care for persons living with Alzheimer's and similar dementia disorders (PLWD). As the number of PLWD rises in the United States from the perhaps 7 million today to possibly 15 million in 2050, the healthcare system will rely on those caregivers even more. It is well established that family caregiving is taxing and stressful and that managing the day-to-day life of PLWD and handling the behavioral and psychological symptoms in dementia (BPSD) that they may exhibit are the main sources of stress. Group-based psychoeducational programs such as the Savvy Caregiver program (SCP) have demonstrated that the acquisition of skills, knowledge, and caregiving mastery can ameliorate caregiving stress - and enhance PLWD quality of life. Many factors, however, preclude caregivers' attendance in group-based programs and limit programs' scalability. To address the issue of access, the researchers have developed the Tele-Savvy program, an online version of SCP that brings groups of caregivers together in facilitator-led synchronous groups and provides substantive educational augmentation through asynchronous e-mail-delivered video lessons.

The first aim of this study is to develop a fully asynchronous online Savvy program that incorporates learning activities that promote both knowledge and skill acquisition and develop and enhance caregivers' felt-sense of caregiving mastery. Developing this education program will utilize input from clinicians, educators, Tele-Savvy facilitators, and caregiver advisors. The second study aim is to determine the feasibility, acceptability and preliminary efficacy of the created online program. This study will recruit 60 family caregivers to take part in a no-control trial of the program. Data will be gathered at baseline, immediately upon course completion and at 3 months post-baseline to assess caregiver distress measures (depression, strain, burden, anxiety), caregiver competence/ mastery, and care recipient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* primary unpaid caregiver for a community-dwelling PLWD
* provide at least 10 hours of direct care per week
* able to read and understand English
* be able to access the course online
* naïve to Savvy or Tele-Savvy

Exclusion Criteria:

* cannot provide consent
* prisoners
* cognitively impaired adult
* not able to clearly understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fayron Epps, PhD, RN, Principal Investigator — Emory University; Carolyn Clevenger, DNP, RN, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be made available for sharing with other researchers, after deidentification.
Supporting Information: Study Protocol
Time Frame: Sharing will begin 3 months and end 5 years following article publication.
Access Criteria: Individual participant data will be made available to researchers who provide a methodologically sound proposal in order to achieve aims in the approved proposal. Proposals should be directed to Dr. Epps at fepps@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Atlanta, USA. Participant enrollment began September 15, 2021 and all follow-up assessments were completed by September 2, 2022.
Groups:
- Fully Asynchronous Online Savvy Program: Family caregivers of a person living with dementia (PLWD) taking part in a fully asynchronous online caregiver education program. The intervention is a fully online, self-administered psychoeducational program designed to enhance caregiver mastery for family and friends providing unpaid care for living with Alzheimer's and similar dementia disorders. Participants are asked to engage with a fully online version of Tele-Savvy for 42 days.
Period: Overall Study
Arm/Group | Fully Asynchronous Online Savvy Program
Started | 60
Completed Month 2 Assessment | 46
Completed Month 3 Assessment | 39
Completed (Completed the study intervention and all study assessments.) | 29
Not Completed | 31
Not completed — Lost to Follow-up | 16
Not completed — Withdrawal by Subject | 5
Not completed — Completed study assessments but did not complete the intervention | 10

BASELINE CHARACTERISTICS:
Groups:
- Fully Asynchronous Online Savvy Program: Family caregivers of PLWD taking part in a fully asynchronous online caregiver education program. The intervention is a fully online, self-administered psychoeducational program designed to enhance caregiver mastery for family and friends providing unpaid care for living with Alzheimer's and similar dementia disorders. Participants are asked to engage with a fully online version of Tele-Savvy for 42 days.
Arm/Group | Fully Asynchronous Online Savvy Program
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.217 (14.438)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 50
  Male | 9
  Non-binary | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 48
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiologic Studies - Depression (CES-D) Score
Description: The CES-D is a 20-item self-report instrument asking respondents if they have experienced symptoms of depression during the past week. Responses are given on a scale of 0 to 3 where "rarely" = 0 and "most of the time" = 3. Total scores range from 0 to 60 and higher scores indicate greater symptoms of depression.
Time Frame: Baseline, Month 2, Month 3
Population: This analysis includes values for the subset of 29 participants who completed the study intervention and the study assessments. Some participants did not complete the study intervention according to study timelines, but they did remain in the study and complete the assessments. In order to report all available data, values are also included for all study participants who completed the survey at the indicated time points, regardless of whether they completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fully Asynchronous Online Savvy Program
Number analyzed (Participants) | 60
score on a scale
  Baseline among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Baseline among those who completed the Online Savvy Program | 11.483 (11.009)
  Month 2 among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Month 2 among those who completed the Online Savvy Program | 9.345 (6.360)
  Month 3 among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Month 3 among those who completed the Online Savvy Program | 8.964 (8.149)
  Baseline among those who completed the survey | 14.317 (11.058)
  Month 2 among those who completed the survey: number analyzed (Participants) | 46
  Month 2 among those who completed the survey | 10.848 (8.200)
  Month 3 among those who completed the survey: number analyzed (Participants) | 39
  Month 3 among those who completed the survey | 10.132 (8.612)

2. Primary Outcome: Zarit Burden Interview Score
Description: The Zarit Burden Interview is a 22-item scale of objective and subjective caregiver burden. Responses are given on a 5-point scale where 0 = never and 4 = nearly always. Total scores range from 0 to 88 where higher scores indicate greater feelings of being burdened with providing care.
Time Frame: Baseline, Month 2, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fully Asynchronous Online Savvy Program
Number analyzed (Participants) | 60
score on a scale
  Baseline among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Baseline among those who completed the Online Savvy Program | 31.207 (12.957)
  Month 2 among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Month 2 among those who completed the Online Savvy Program | 29.138 (10.395)
  Month 3 among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Month 3 among those who completed the Online Savvy Program | 26.296 (9.474)
  Baseline among those who completed the survey | 35.050 (14.274)
  Month 2 among those who completed the survey: number analyzed (Participants) | 46
  Month 2 among those who completed the survey | 31.239 (10.754)
  Month 3 among those who completed the survey: number analyzed (Participants) | 39
  Month 3 among those who completed the survey | 28.730 (10.235)

3. Primary Outcome: State-Trait Anxiety Inventory (STAI) Score
Description: The STAI is a 20-item self-report scale of positive and negative anxiety experiences. Responses are given on a 4-point scale where 1 = not at all and 4 = very much so. Total scores range from 20 to 80 and higher scores indicate greater anxiety.
Time Frame: Baseline, Month 2, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fully Asynchronous Online Savvy Program
Number analyzed (Participants) | 60
score on a scale
  Baseline among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Baseline among those who completed the Online Savvy Program | 31.793 (9.777)
  Month 2 among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Month 2 among those who completed the Online Savvy Program | 31.793 (8.104)
  Month 3 among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Month 3 among those who completed the Online Savvy Program | 29.893 (8.230)
  Baseline among those who completed the survey | 34.862 (11.190)
  Month 2 among those who completed the survey: number analyzed (Participants) | 46
  Month 2 among those who completed the survey | 31.761 (9.053)
  Month 3 among those who completed the survey: number analyzed (Participants) | 39
  Month 3 among those who completed the survey | 31.103 (9.167)

4. Primary Outcome: Caregiver Mastery Scale - Caregiving Competence Score
Description: The Caregiving Mastery instrument assesses caregiver mastery of 3 different realms of caregiving situations: Relational Deprivation, Caregiving Competence, and Management of Situation. The Caregiving Competence subscale asks caregivers about their thoughts about the caregiving they provide with 4 items where responses are given on a 4-point scale where "not at all" = 1 and "completely" or "very" = 4. Total scores range from 4 to 16 where higher scores indicate greater feelings of competence with caregiving.
Time Frame: Baseline, Month 2, Month 3
Population: Participants with incomplete responses were removed from this analysis. Of the 29 participants who completed the study intervention and assessments, 4 had missing responses for this survey at any time point, resulting in 25 participants analyzed. Values are also included for all study participants responding to surveys at the indicated time points, even if they did not complete the intervention; of these 8 had missing responses on this survey at Baseline and 1 had missing responses at Month 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fully Asynchronous Online Savvy Program
Number analyzed (Participants) | 52
score on a scale
  Baseline among those who completed the Online Savvy Program: number analyzed (Participants) | 25
  Baseline among those who completed the Online Savvy Program | 12.160 (1.700)
  Month 2 among those who completed the Online Savvy Program: number analyzed (Participants) | 25
  Month 2 among those who completed the Online Savvy Program | 12.821 (1.945)
  Month 3 among those who completed the Online Savvy Program: number analyzed (Participants) | 25
  Month 3 among those who completed the Online Savvy Program | 13.143 (2.085)
  Baseline among those who completed the survey | 11.481 (2.330)
  Month 2 among those who completed the survey: number analyzed (Participants) | 45
  Month 2 among those who completed the survey | 12.689 (1.998)
  Month 3 among those who completed the survey: number analyzed (Participants) | 39
  Month 3 among those who completed the survey | 13.026 (2.146)

5. Primary Outcome: Revised Memory and Behavior Problem Checklist (RMBPC) Frequency Score
Description: The RMBPC is a 24-item scale reporting on frequency of disturbing care recipient behaviors and severity or caregiver reactions to these behaviors. Respondents indicate how frequently problems have occurred on a 5-point scale where 0 = never occurred and 4 = daily or more often. Total frequency scores range from 0 to 96 with higher scores indicating greater frequency of memory and behavior problems exhibited by the PLWD.
Time Frame: Baseline, Month 2, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fully Asynchronous Online Savvy Program
Number analyzed (Participants) | 60
score on a scale
  Baseline among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Baseline among those who completed the Online Savvy Program | 40.276 (12.015)
  Month 2 among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Month 2 among those who completed the Online Savvy Program | 36.345 (9.529)
  Month 3 among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Month 3 among those who completed the Online Savvy Program | 34.786 (9.796)
  Baseline among those who completed the survey | 40.407 (13.849)
  Month 2 among those who completed the survey: number analyzed (Participants) | 46
  Month 2 among those who completed the survey | 35.739 (10.784)
  Month 3 among those who completed the survey: number analyzed (Participants) | 39
  Month 3 among those who completed the survey | 34.897 (9.784)

6. Primary Outcome: Revised Memory and Behavior Problem Checklist (RMBPC) Reaction Score
Description: The RMBPC is a 24-item scale reporting on frequency of disturbing care recipient behaviors and severity or caregiver reactions to these behaviors. Respondents indicate the degree to which problems have bothered or upset them on a 5-point scale where 0 = not at all and 4 = extremely. Total reaction scores range from 0 to 96 with higher scores indicating more bothered or upset by memory and behavior problems exhibited by the PLWD.
Time Frame: Baseline, Month 2, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fully Asynchronous Online Savvy Program
Number analyzed (Participants) | 60
score on a scale
  Baseline among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Baseline among those who completed the Online Savvy Program | 18.483 (10.534)
  Month 2 among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Month 2 among those who completed the Online Savvy Program | 12.828 (7.016)
  Month 3 among those who completed the Online Savvy Program: number analyzed (Participants) | 29
  Month 3 among those who completed the Online Savvy Program | 12.893 (7.420)
  Baseline among those who completed the survey | 20.167 (12.238)
  Month 2 among those who completed the survey: number analyzed (Participants) | 46
  Month 2 among those who completed the survey | 12.522 (7.453)
  Month 3 among those who completed the survey: number analyzed (Participants) | 39
  Month 3 among those who completed the survey | 13.132 (7.977)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning when consent was given to participant in the study and continued through the final assessment at Month 3.
Arm/Group | Fully Asynchronous Online Savvy Program
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT04951037/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT04951037/ICF_001.pdf